CLINICAL TRIAL: NCT05839860
Title: The Effect of Low and High Salt Intake on Hydration Status and Gastrointestinal Discomfort During Seven Hours of Dry Fasting
Brief Title: Salt Intake, Hydration Status and Gastrointestinal Discomfort During Fasting
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oxford Brookes University (Other)
Responsible Party: Principal Investigator, Dr. Sangeetha Thondre, Senior Lecturer, Oxford Brookes University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: UREC 221630
Record Dates: First submitted 2023-03-23; First posted 2023-05-03 (Actual); Last update posted 2023-09-06 (Actual); Status verified 2023-09

CONDITIONS: Healthy
MeSH Terms: interventions — Salts

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 3 g salt (Placebo Comparator): Tomatoes with 3 g salt
  Interventions: Other: Salt 3 g
- 6 g salt (Experimental): Tomatoes with 6 g salt and 1 L of water
  Interventions: Other: Salt 6 g
- 9 g salt (Experimental): Tomatoes with 9 g salt and 1 L of water
  Interventions: Other: Salt 9 g

INTERVENTIONS:
Other: Salt 3 g — Placebo group taking a breakfast meal and 3g salt on tomatoes before fasting for 7 hours
  Arms: 3 g salt
Other: Salt 6 g — Intervention group taking a breakfast meal and 6g salt on tomatoes plus 1 L water before fasting for 7 hours
  Arms: 6 g salt
Other: Salt 9 g — Intervention group taking a breakfast meal and 9g salt on tomatoes plus 1 L water before fasting for 7 hours
  Arms: 9 g salt

SUMMARY:
This study is part of a hyperhydration project and it has been designed based on a scoping review (Hyperhydration in healthy adults: a scoping review on different methodologies and vehicles utilized) and a previous study (Dietary patterns and gastrointestinal discomfort during Ramadan in a UK Muslim population). The current study aims to examine the impact of different levels of salt intake (6 & 9 grams) with [15 milliliters per kilogram of bodyweight (ml/ kg/ bw)] of water intake during 7 hours of dry fasting compared to a control group (3g salt) under the state of water balance (euhydrated). A previous study and a review by the authors highlighted the potential negative impact of salt and fasting on gastrointestinal (GI) discomfort; hence, the potential negative side effects on gastrointestinal (GI) discomfort during the intervention period will be investigated. By studying a hyperhydration protocol, this research will help the population to reduce dehydration during dry fasting. By doing so, it may improve the quality of life during Ramadan fasting.

DETAILED DESCRIPTION:
Dry fasting has been reported to cause changes in body weight, lipid profile, blood pressure, glucose level, metabolism, hormones homeostasis, and hydration status. A scoping review by the investigators highlighted that dehydration had been linked to changes in plasma volume and osmolality (concentration of all chemical particles), urine volume and osmolality, blood pressure, glucocorticoid hormones, body weight loss, negative impact on mood, irritability, short-term memory, and work productivity. It has been reported that prolonged dry fasting can contribute to a loss of up to 1.5 kg in body weight on the day after fasting. This weight loss is associated with loss of body water.

Hyperhydration (overhydration) has not yet been defined. However, any improvement in the fluid matrix in the plasma volume is considered hyperhydration. Simulating hyperhydration strategies, such as those used by athletes competing in long-distance events and in hot environments, has the potential to reduce the level of dehydration during dry fasting.

Sodium and water intake have essential roles in maintaining and improving the fluid matrix in plasma. By investigating the relationship between sodium and water intake on biomarkers such as urine sodium concentration, blood pressure, speed of urine production, urine colour, urine specific gravity, and net body fluid balance, it is possible to distinguish the impact of hyperhydration protocols on hydration levels.

The primary aim of this study is to examine the impact of salt intake (6 & 9 g/l) on the level of hydration by measuring urine sodium, urine potassium, urine production, and changes in body weight compared to the control group during 8 hours of dry fasting. The secondary outcome of this study will be the impact of the hyperhydration protocol on GI discomfort.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 to 45
* BMI between 18.5 and 29.9
* No higher (140/90mmHg) or lower (80/60mmHg) blood pressure
* Non-pregnant or lactating
* No diabetes (type 1 & 2)
* No gastrointestinal disease such as inflammatory bowel disease (IBD) or Irritable bowel syndrome (IBS)
* No disease including the common cold and high cholesterol (total cholesterol above 5 mmol/l)
* No covid symptoms
* No allergy to the food in the meal list and tomatoes

Exclusion Criteria:

* Aged <18 or >45 years
* BMI between <18.5 or > 29.9
* Higher (>140/90mmHg) or lower (<80/60mmHg) blood pressure
* Pregnant or lactating
* Having diabetes (type 1 & 2)
* Having gastrointestinal disease such as inflammatory bowel disease (IBD) or Irritable bowel syndrome (IBS)
* Having disease including the common cold and high cholesterol (total cholesterol above 5 mmol/l)
* Having covid symptoms
* Having allergy to the food in the meal list and tomatoes

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 23 (Actual)
Dates: Start 2023-02-14 (Actual); Primary Completion 2023-05-31 (Actual); Study Completion 2023-07-31 (Actual)

PRIMARY OUTCOMES:
Total urine production baseline | 0 hour
  Volume of urine produced at baseline
Total urine production 1 hour | 1 hour
  Volume of urine produced at 1 hour after starting fasting
Total urine production 2 hours | 2 hours
  Volume of urine produced at at 2 hours after starting fasting
Total urine production 3 hours | 3 hours
  Volume of urine produced at at 3 hours after starting fasting
Total urine production 4 hours | 4 hours
  Volume of urine produced at at 4 hours after starting fasting
Total urine production 5 hours | 5 hours
  Volume of urine produced at at 5 hours after starting fasting
Total urine production 6 hours | 6 hours
  Volume of urine produced at at 6 hours after starting fasting
Total urine production 7 hours | 7 hours
  Volume of urine produced at at 7 hours after starting fasting
Body weight baseline | 0 hours
  Body weight at baseline before fasting
Body weight 1 hour | 1 hour
  Body weight at 1 hour after starting fasting
Body weight 2 hours | 2 hours
  Body weight at 2 hours after starting fasting
Body weight 3 hours | 3 hours
  Body weight at 3 hours after starting fasting
Body weight 4 hours | 4 hours
  Body weight at 4 hours after starting fasting
Body weight 5 hours | 5 hours
  Body weight at 5 hours after starting fasting
Body weight 6 hours | 6 hours
  Body weight at 6 hours after starting fasting
Body weight 7 hours | 7 hours
  Body weight at 7 hours after starting fasting
Urinary sodium baseline | 0 hours
  Urinary sodium at baseline before starting fasting
Urinary sodium 1 hour | 1 hour
  Urinary sodium at 1 hour after starting fasting
Urinary sodium 2 hours | 2 hours
  Urinary sodium at 2 hours after starting fasting
Urinary sodium 3 hours | 3 hours
  Urinary sodium at 3 hours after starting fasting
Urinary sodium 4 hours | 4 hours
  Urinary sodium at 4 hours after starting fasting
Urinary sodium 5 hours | 5 hours
  Urinary sodium at 5 hours after starting fasting
Urinary sodium 6 hours | 6 hours
  Urinary sodium at 6 hours after starting fasting
Urinary sodium 7 hours | 7 hours
  Urinary sodium at 7 hours after starting fasting
Urinary potassium baseline | 0 hours
  Urinary potassium at baseline before starting fasting
Urinary potassium 1 hour | 1 hour
  Urinary potassium at 1 hour after starting fasting
Urinary potassium 2 hours | 2 hours
  Urinary potassium at 2 hours after starting fasting
Urinary potassium 3 hours | 3 hours
  Urinary potassium at 3 hours after starting fasting
Urinary potassium 4 hours | 4 hours
  Urinary potassium at 4 hours after starting fasting
Urinary potassium 5 hours | 5 hours
  Urinary potassium at 5 hours after starting fasting
Urinary potassium 6 hours | 6 hours
  Urinary potassium at 6 hours after starting fasting
Urinary potassium 7 hours | 7 hours
  Urinary potassium at 7 hours after starting fasting
Urine colour baseline | 0 hours
  Urine colour at baseline before starting fasting
Urine colour 1 hour | 1 hour
  Urine colour at 1 hour after starting fasting
Urine colour 2 hours | 2 hours
  Urine colour at 2 hours after starting fasting
Urine colour 3 hours | 3 hours
  Urine colour at 3 hours after starting fasting
Urine colour 4 hours | 4 hours
  Urine colour at 4 hours after starting fasting
Urine colour 5 hours | 5 hours
  Urine colour at 5 hours after starting fasting
Urine colour 6 hours | 6 hours
  Urine colour at 6 hours after starting fasting
Urine colour 7 hours | 7 hours
  Urine colour at 7 hours after starting fasting
Urine specific gravity baseline | 0 hours
  Urine specific gravity at baseline before starting fasting
Urine specific gravity 1 hour | 1 hour
  Urine specific gravity at 1 hour after starting fasting
Urine specific gravity 2 hours | 2 hours
  Urine specific gravity at 2 hours after starting fasting
Urine specific gravity 3 hours | 3 hours
  Urine specific gravity at 3 hours after starting fasting
Urine specific gravity 4 hours | 4 hours
  Urine specific gravity at 4 hours after starting fasting
Urine specific gravity 5 hours | 5 hours
  Urine specific gravity at 5 hours after starting fasting
Urine specific gravity 6 hours | 6 hours
  Urine specific gravity at 6 hours after starting fasting
Urine specific gravity 7 hours | 7 hours
  Urine specific gravity at 7 hours after starting fasting

SECONDARY OUTCOMES:
Gastrointestinal discomfort baseline | 0 hours
  Gastrointestinal discomfort at baseline before starting fasting using a Gastrointestinal Symptoms Questionnaire to measure 1.Abdominal pain 2.Epigastric pain (pain or discomfort right below your ribs in the area of your upper abdomen) 3. Heartburn 4. Regurgitation 5. Abdominal rumbling 6. Bloating 7. Empty feeling 8. Nausea 9. Vomiting 10. Loss of appetite 11. Postprandial fullness (an unpleasant sensation like prolonged persistence of food in the stomach) 12. belching (otherwise known as burping or eructation) 13. Flatulence (buildup of gas in the digestive system that can lead to abdominal discomfort) on a 7 point scale labelled 0 for none, 1 for mild, 2 for moderate, 3 for quite a lot, 4 for severe, 5 for very severe, 6 for unbearable. Higher scores mean worst outcome.
Gastrointestinal discomfort 1 hour | 1 hour
  Gastrointestinal discomfort at 1 hour after starting fasting using a Gastrointestinal Symptoms Questionnaire to measure 1.Abdominal pain 2.Epigastric pain (pain or discomfort right below your ribs in the area of your upper abdomen) 3. Heartburn 4. Regurgitation 5. Abdominal rumbling 6. Bloating 7. Empty feeling 8. Nausea 9. Vomiting 10. Loss of appetite 11. Postprandial fullness (an unpleasant sensation like prolonged persistence of food in the stomach) 12. belching (otherwise known as burping or eructation) 13. Flatulence (buildup of gas in the digestive system that can lead to abdominal discomfort) on a 7 point scale labelled 0 for none, 1 for mild, 2 for moderate, 3 for quite a lot, 4 for severe, 5 for very severe, 6 for unbearable. Higher scores mean worst outcome.
Gastrointestinal discomfort 2 hours | 2 hours
  Gastrointestinal discomfort at 2 hours after starting fasting using a Gastrointestinal Symptoms Questionnaire to measure 1.Abdominal pain 2.Epigastric pain (pain or discomfort right below your ribs in the area of your upper abdomen) 3. Heartburn 4. Regurgitation 5. Abdominal rumbling 6. Bloating 7. Empty feeling 8. Nausea 9. Vomiting 10. Loss of appetite 11. Postprandial fullness (an unpleasant sensation like prolonged persistence of food in the stomach) 12. belching (otherwise known as burping or eructation) 13. Flatulence (buildup of gas in the digestive system that can lead to abdominal discomfort) on a 7 point scale labelled 0 for none, 1 for mild, 2 for moderate, 3 for quite a lot, 4 for severe, 5 for very severe, 6 for unbearable. Higher scores mean worst outcome.
Gastrointestinal discomfort 3 hours | 3 hours
  Gastrointestinal discomfort at 3 hours after starting fasting using a Gastrointestinal Symptoms Questionnaire to measure 1.Abdominal pain 2.Epigastric pain (pain or discomfort right below your ribs in the area of your upper abdomen) 3. Heartburn 4. Regurgitation 5. Abdominal rumbling 6. Bloating 7. Empty feeling 8. Nausea 9. Vomiting 10. Loss of appetite 11. Postprandial fullness (an unpleasant sensation like prolonged persistence of food in the stomach) 12. belching (otherwise known as burping or eructation) 13. Flatulence (buildup of gas in the digestive system that can lead to abdominal discomfort) on a 7 point scale labelled 0 for none, 1 for mild, 2 for moderate, 3 for quite a lot, 4 for severe, 5 for very severe, 6 for unbearable. Higher scores mean worst outcome.
Gastrointestinal discomfort 4 hours | 4 hours
  Gastrointestinal discomfort at 4 hours after starting fasting using a Gastrointestinal Symptoms Questionnaire to measure 1.Abdominal pain 2.Epigastric pain (pain or discomfort right below your ribs in the area of your upper abdomen) 3. Heartburn 4. Regurgitation 5. Abdominal rumbling 6. Bloating 7. Empty feeling 8. Nausea 9. Vomiting 10. Loss of appetite 11. Postprandial fullness (an unpleasant sensation like prolonged persistence of food in the stomach) 12. belching (otherwise known as burping or eructation) 13. Flatulence (buildup of gas in the digestive system that can lead to abdominal discomfort) on a 7 point scale labelled 0 for none, 1 for mild, 2 for moderate, 3 for quite a lot, 4 for severe, 5 for very severe, 6 for unbearable. Higher scores mean worst outcome.
Gastrointestinal discomfort 5 hours | 5 hours
  Gastrointestinal discomfort at 5 hours after starting fasting using a Gastrointestinal Symptoms Questionnaire to measure 1.Abdominal pain 2.Epigastric pain (pain or discomfort right below your ribs in the area of your upper abdomen) 3. Heartburn 4. Regurgitation 5. Abdominal rumbling 6. Bloating 7. Empty feeling 8. Nausea 9. Vomiting 10. Loss of appetite 11. Postprandial fullness (an unpleasant sensation like prolonged persistence of food in the stomach) 12. belching (otherwise known as burping or eructation) 13. Flatulence (buildup of gas in the digestive system that can lead to abdominal discomfort) on a 7 point scale labelled 0 for none, 1 for mild, 2 for moderate, 3 for quite a lot, 4 for severe, 5 for very severe, 6 for unbearable. Higher scores mean worst outcome.
Gastrointestinal discomfort 6 hours | 6 hours
  Gastrointestinal discomfort at 6 hours after starting fasting using a Gastrointestinal Symptoms Questionnaire to measure 1.Abdominal pain 2.Epigastric pain (pain or discomfort right below your ribs in the area of your upper abdomen) 3. Heartburn 4. Regurgitation 5. Abdominal rumbling 6. Bloating 7. Empty feeling 8. Nausea 9. Vomiting 10. Loss of appetite 11. Postprandial fullness (an unpleasant sensation like prolonged persistence of food in the stomach) 12. belching (otherwise known as burping or eructation) 13. Flatulence (buildup of gas in the digestive system that can lead to abdominal discomfort) on a 7 point scale labelled 0 for none, 1 for mild, 2 for moderate, 3 for quite a lot, 4 for severe, 5 for very severe, 6 for unbearable. Higher scores mean worst outcome.
Gastrointestinal discomfort 7 hours | 7 hours
  Gastrointestinal discomfort at 7 hours after starting fasting using a Gastrointestinal Symptoms Questionnaire to measure 1.Abdominal pain 2.Epigastric pain (pain or discomfort right below your ribs in the area of your upper abdomen) 3. Heartburn 4. Regurgitation 5. Abdominal rumbling 6. Bloating 7. Empty feeling 8. Nausea 9. Vomiting 10. Loss of appetite 11. Postprandial fullness (an unpleasant sensation like prolonged persistence of food in the stomach) 12. belching (otherwise known as burping or eructation) 13. Flatulence (buildup of gas in the digestive system that can lead to abdominal discomfort) on a 7 point scale labelled 0 for none, 1 for mild, 2 for moderate, 3 for quite a lot, 4 for severe, 5 for very severe, 6 for unbearable. Higher scores mean worst outcome.
Blood Pressure baseline | 0 hours
  Systolic and Diastolic Blood Pressure at baseline before starting fasting
Blood Pressure 1 hour | 1 hour
  Systolic and Diastolic Blood Pressure at 1 hour after starting fasting
Blood Pressure 2 hours | 2 hours
  Systolic and Diastolic Blood Pressure at 2 hours after starting fasting
Blood Pressure 3 hours | 3 hours
  Systolic and Diastolic Blood Pressure at 3 hours after starting fasting
Blood Pressure 4 hours | 4 hours
  Systolic and Diastolic Blood Pressure at 4 hours after starting fasting
Blood Pressure 5 hours | 5 hours
  Systolic and Diastolic Blood Pressure at 5 hours after starting fasting
Blood Pressure 6 hours | 6 hours
  Systolic and Diastolic Blood Pressure at 6 hours after starting fasting
Blood Pressure 7 hours | 7 hours
  Systolic and Diastolic Blood Pressure at 7 hours after starting fasting
Perception of thirst at baseline | 0 hours
  Perception of thirst at baseline before starting fasting using a 7 point scale labelled as 1=not thirsty at all, 2=not thirsty, 3=not very thirsty, 4=neutral, 5=thirsty, 6=very thirsty and 7=very, very thirsty.
Perception of thirst at 1 hour | 1 hour
  Perception of thirst at 1 hour after starting fasting using a 7 point scale labelled as 1=not thirsty at all, 2=not thirsty, 3=not very thirsty, 4=neutral, 5=thirsty, 6=very thirsty and 7=very, very thirsty.
Perception of thirst at 2 hours | 2 hours
  Perception of thirst at 2 hours after starting fasting using a 7 point scale labelled as 1=not thirsty at all, 2=not thirsty, 3=not very thirsty, 4=neutral, 5=thirsty, 6=very thirsty and 7=very, very thirsty.
Perception of thirst at 3 hours | 3 hours
  Perception of thirst at 3 hours after starting fasting using a 7 point scale labelled as 1=not thirsty at all, 2=not thirsty, 3=not very thirsty, 4=neutral, 5=thirsty, 6=very thirsty and 7=very, very thirsty.
Perception of thirst at 4 hours | 4 hours
  Perception of thirst at 4 hours after starting fasting using a 7 point scale labelled as 1=not thirsty at all, 2=not thirsty, 3=not very thirsty, 4=neutral, 5=thirsty, 6=very thirsty and 7=very, very thirsty.
Perception of thirst at 5 hours | 5 hours
  Perception of thirst at 5 hours after starting fasting using a 7 point scale labelled as 1=not thirsty at all, 2=not thirsty, 3=not very thirsty, 4=neutral, 5=thirsty, 6=very thirsty and 7=very, very thirsty.
Perception of thirst at 6 hours | 6 hours
  Perception of thirst at 6 hours after starting fasting using a 7 point scale labelled as 1=not thirsty at all, 2=not thirsty, 3=not very thirsty, 4=neutral, 5=thirsty, 6=very thirsty and 7=very, very thirsty.
Perception of thirst at 7 hours | 7 hours
  Perception of thirst at 7 hours after starting fasting using a 7 point scale labelled as 1=not thirsty at all, 2=not thirsty, 3=not very thirsty, 4=neutral, 5=thirsty, 6=very thirsty and 7=very, very thirsty.

CONTACTS AND LOCATIONS:
Overall Officials: Sangeetha Thondre, PhD, Principal Investigator — Oxford Brookes University
Locations (1):
- Oxford Brookes Centre for Nutrition and Health, Oxford, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Goulet EDB, De La Flore A, Savoie FA, Gosselin J. Salt + Glycerol-Induced Hyperhydration Enhances Fluid Retention More Than Salt- or Glycerol-Induced Hyperhydration. Int J Sport Nutr Exerc Metab. 2018 May 1;28(3):246-252. doi: 10.1123/ijsnem.2017-0310. Epub 2018 May 17. PMID 29140136
- [Background] Zanetti D, Bergman H, Burgess S, Assimes TL, Bhalla V, Ingelsson E. Urinary Albumin, Sodium, and Potassium and Cardiovascular Outcomes in the UK Biobank: Observational and Mendelian Randomization Analyses. Hypertension. 2020 Mar;75(3):714-722. doi: 10.1161/HYPERTENSIONAHA.119.14028. Epub 2020 Feb 3. PMID 32008434